CLINICAL TRIAL: NCT05452759
Title: Randomized Controlled Trial of Spiral Exhalation Device Oxygen Therapy to Improve the Treatment Effect of Patients With Severe Pneumonia.
Brief Title: Research of Spiral Exhalation Device Oxygen Therapy to Improve the Treatment Effect of Patients With Severe Pneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20223357002
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- new type of tracheotomy high-flow oxygen therapy (NTHF) (Experimental): Using NTHF, adjust the MR850 humidifier to invasive automatic gear, the temperature sensor automatically adjusts and maintains the gas temperature at the entrance of the tracheal tube at 37°C according to the feedback temperature, and monitors and maintains SpO2 between 94% and 100%. The monitored pulse oxygen saturation (SpO2) is used to adjust the concentration of the venturi valve and the corresponding oxygen flow rate. At the preset gas flow rate levels of 40L/min, 50L/min and 60L/min, the test pipeline is connected to optimize the breath. The actual gas flow rate value and the gas flow rate loss difference before and after the gas joint (screw joint), and at the corresponding gas flow rate, measure the gas temperature and humidity at the near-patient end of the pipeline.
  Interventions: Device: high-flow oxygen therapy device for Severe pneumonia patients with artificial airway
- Respiratory Humidification Treatment（ AIRVO TM 2） (Active Comparator): Use AIRVOTM2 (Fisher & Paykel, Auckland, New Zealand), select the output gas temperature of 37°C, monitor and maintain SpO2 between 94% and 100%, and adjust the output gas flow rate of the therapy device to 40L/min, 50L/min and 60L/min, respectively. min, measure the actual gas flow rate value and the gas flow rate loss difference before and after each flow rate horizontal pipeline is connected to the conventional exhalation joint (matching special exhalation joint), and measure the gas temperature and humidity near the patient end of the pipeline at the corresponding gas flow rate.
  Interventions: Device: AIRVOTM2 device for Severe pneumonia patients with artificial airway

INTERVENTIONS:
Device: high-flow oxygen therapy device for Severe pneumonia patients with artificial airway — Using NTHF, adjust the MR850 humidifier to invasive automatic gear, the temperature sensor automatically adjusts and maintains the gas temperature at the entrance of the tracheal tube at 37°C according to the feedback temperature, and monitors and maintains SpO2 between 94% and 100%. The monitored pulse oxygen saturation (SpO2) is used to adjust the concentration of the venturi valve and the corresponding oxygen flow rate. At the preset gas flow rate levels of 40L/min, 50L/min and 60L/min, the test pipeline is connected to optimize the breath. The actual gas flow rate value and the gas flow rate loss difference before and after the gas joint (screw joint), and at the corresponding gas flow rate, measure the gas temperature and humidity at the near-patient end of the pipeline.
  Arms: new type of tracheotomy high-flow oxygen therapy (NTHF)
Device: AIRVOTM2 device for Severe pneumonia patients with artificial airway — Use AIRVOTM2 (Fisher & Paykel, Auckland, New Zealand), select the output gas temperature of 37°C, monitor and maintain SpO2 between 94% and 100%, and adjust the output gas flow rate of the therapy device to 40L/min, 50L/min and 60L/min, respectively. min, measure the actual gas flow rate value and the gas flow rate loss difference before and after each flow rate horizontal pipeline is connected to the conventional exhalation joint (matching special exhalation joint), and measure the gas temperature and humidity near the patient end of the pipeline at the corresponding gas flow rate.
  Arms: Respiratory Humidification Treatment（ AIRVO TM 2）

SUMMARY:
Severe pneumonia has a high morbidity and mortality. Humidified oxygen therapy, mechanical ventilation, and removal of airway secretions are the main non-drug treatments. However, mechanical ventilation leads to a high economic burden, and ventilator-associated pneumonia may increase patient mortality. Therefore, it is necessary to conduct in-depth research on early release from the ventilator and oxygen therapy. Studies have shown that high-flow nasal oxygen therapy (HFNC) improves airway humidification and oxygenation in patients. The respiratory humidification therapy device (AIRVOTM2) is mainly used internationally, but clinical studies on artificial airway patients are limited.

In the previous study, we improved the "New Artificial Airway High Flow Humidification Oxygen Therapy Device" (NTHF) to improve the accuracy of gas flow rate, and unified the baseline with AIRVOTM2. The status quo of the obvious differences in the airway humidification effect of patients. The pre-experiment again found that the gas flow rate consumption was significantly lower than that of AIRVOTM2 after the NTHF exhalation port was optimized, and the gas flow rate was proportional to the inhaled gas humidity. Based on this, we hypothesized that the flow rate of the optimized expiratory port of NTHF is more stable than that of AIRVOTM2, which can improve the airway humidification effect of patients. We intend to adopt a randomized controlled clinical study design, by comparing the application of two oxygen therapy devices in patients with severe pneumonia artificial airway, to explore whether NTHF can promote the clearance of airway secretions in patients with severe pneumonia and improve the therapeutic effect of severe pneumonia. Oxygen therapy nursing mode in patients with severe pneumonia artificial airway.

DETAILED DESCRIPTION:
On the basis of the previous study, through the randomized controlled study design, it is proved that the spiral oxygen therapy exhalation port can reduce the consumption of the gas flow rate of the oxygen therapy device, improve the airway humidification and defense system ability of patients, and promote the infection control of patients with severe pneumonia. Innovate the oxygen therapy mode of NTHF in artificial airway patients with severe pneumonia to achieve the purpose of reducing mechanical ventilation and improving the therapeutic effect.

Before the start of the study, all enrolled patients were required to sign an informed consent form. Patients who met the inclusion criteria were divided into NTHF exhalation port optimization group (experimental group) and AIRVOTM2 exhalation port conventional group (control group) according to the ratio of 1:1, with 78 cases in each group. The method of block randomization with random block size is adopted, and the random number and grouping result generated by the computer are used to make a random grouping card, which is stored in a sealed and opaque envelope with the same surface. And the envelopes are numbered one-time according to the sequence number of the random grouping method. The researcher selects the corresponding envelope according to the order in which the subjects entered the experiment, obtains the grouping number, and gives the subjects different high-flow humidified oxygen therapy strictly according to the card.

Blind method: This study is a single-blind study. The researcher clearly defines the treatment group, but the index evaluation, data collection and data statistics are completed by different trained researchers, and the treatment group is not clear.

Intervention group: use NTHF, adjust the MR850 humidifier to invasive automatic gear, the temperature sensor automatically adjusts and maintains the gas temperature at the entrance of the tracheal tube at 37°C according to the feedback temperature, and monitors and maintains SpO2 between 94% and 100%. , adjust the concentration of the venturi valve and the corresponding oxygen flow according to the monitored pulse oxygen saturation (SpO2), and test the pipeline at the preset gas flow rate levels of 40L/min, 50L/min and 60L/min respectively. Connect the actual gas flow rate value and gas flow rate loss difference before and after the optimized expiratory joint (screw joint), and measure the gas temperature and humidity at the near-patient end of the pipeline at the corresponding gas flow rate.

Control group: use AIRVOTM2 (Fisher & Paykel, Auckland, New Zealand), select the output gas temperature of 37°C, monitor and maintain SpO2 between 94% and 100%, and adjust the output gas flow rate of the therapeutic apparatus to 40L/min and 50L/min respectively. and 60L/min, measure the actual gas flow rate and the gas flow loss difference before and after each flow rate horizontal pipeline is connected to the conventional exhalation joint (matching special exhalation joint), and at the corresponding gas flow rate, measure the gas near the patient end of the pipeline. temperature and humidity.

ELIGIBILITY:
Inclusion Criteria:

* The age of the patient is ≥18 years old and meets the diagnostic criteria for severe pneumonia.

  * The patient has artificial airway preparation or has been released from the ventilator.

    * Needs to receive oxygen therapy for more than 24 hours.

      * The expected retention days of the tracheal tube ≥ 7 days ⑤ Sign the informed consent

Exclusion Criteria:

* Patients with one-lung ventilation

  * Patients with pregnancy and end-stage tumors ③Airway hemorrhage

    * Medical history of airway injury, pulmonary trauma, lung surgery ⑤ Hypothermia (<35℃), restrictive body fluid deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
level of flow rate proximal to the patient | On the day of using the high-flow humidified oxygen therapy device
  The gas flow rate was measured using the MF5612 split display gas mass flowmeter produced by Sixiang Microelectronics in the United States
level of flow rate proximal to the patient | 48 hours after start of high flow oxygen therapy
  The gas flow rate was measured using the MF5612 split display gas mass flowmeter produced by Sixiang Microelectronics in the United States
level of flow rate proximal to the patient | 7th days after start of high flow oxygen therapy
  The gas flow rate was measured using the MF5612 split display gas mass flowmeter produced by Sixiang Microelectronics in the United States

SECONDARY OUTCOMES:
level of sputum viscosity | 24th, 48th and 7th days after start of high flow oxygen therapy
  sputum viscosity is assessed with a sputum viscometer
Level of oxygenation | 24th, 48th and 7th days after start of high flow oxygen therapy
  Oxygenation is assessed by arterial blood gas sample

OTHER OUTCOMES:
Patient satisfaction scoreg greater than or equal to 90 | the 7th day after start of high flow oxygen therapy
  Using Hospital Designated Satisfaction Questionnaire which include comfort, bloating, dry mouth, ability to hear and speak（Total score is 100 points）

CONTACTS AND LOCATIONS:
Overall Officials: MEI YANGMEI, Study Chair — Shenzhen Second People's Hospital
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No